CLINICAL TRIAL: NCT03696823
Title: Assessment of Routine Use of Critical View of Safety in Laparoscopic Cholecystectomy, Prospective Cohort Study
Brief Title: Critical View of Safety in Laparoscopic Cholecystectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abanoub Khalf Henry Romany, principal investigator, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: laparoscopic cholecystectomy
Record Dates: First submitted 2018-09-20; First posted 2018-10-05 (Actual); Last update posted 2018-10-05 (Actual); Status verified 2018-10

CONDITIONS: Chronic Calculous Cholecystitis
MeSH Terms: interventions — Cholecystectomy, Laparoscopic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: laparoscopic cholecystectomy — treatment of chronic calcular cholecystitis laparoscopically

SUMMARY:
This prospective cohort study aims to assess feasibility and safety of the approach of critical view of safety during laparoscopic cholecystectomy

DETAILED DESCRIPTION:
Since the introduction and routine use of laparoscopic cholecystectomy in the 1990s, the reported incidence of biliary injuries has doubled to 0.4%.

Many factors have been shown to influence the risk of biliary injury including patient factors (obesity, older age, male gender and adhesions), local factors (severe gallbladder inflammation/infection, aberrant anatomy and haemorrhage) as well as surgeon experience.

Identifying the common bile duct as the cystic duct is the commonest cause of major bile duct injury Active identification of cystic structures within Calot's triangle is the key to a reduction in biliary injury. Strasberg first coined the term 'critical view of safety' (CVS) in 1958 and this approach of identification of cystic structures has been adopted by many surgeons as the standard of operative technique to reduce the incidence of biliary injury.

To fulfil the criteria for a CVS requires Calot's triangle to be cleared free of fat and fibrous tissue ('fat cleared'), for the lowest part of the gallbladder to be dissected free from the cystic plate ('liver visible') and for there to be only two structures entering the gallbladder ('2 structures').

The published rate of bile duct injury with this approach is very low However more studies are needed to assess risk benefit rate of this approach.

ELIGIBILITY:
Inclusion Criteria:

* include all patients who will have laparoscopic cholecystectomy

Exclusion Criteria :-

* Emergency laparoscopic cholecystectomy
* Liver cirrhosis
* HCV & HBV

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-10-01 (Estimated); Primary Completion 2019-10 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
(CVS) is a mean of target identification, the targets being the cystic duct and artery for changes in the incidence of biliary injury. Identifying the common bile duct as the cystic duct is the commonest cause of major bile duct injury. | baseline & 6 months
  Identifying the common bile duct as the cystic duct is the commonest cause of major bile duct injury.
  Active identification of cystic structures within Calot's triangle is the key to a reduction in biliary injury.
  To fulfil the criteria for a CVS requires Calot's triangle to be cleared free of fat and fibrous tissue ('fat cleared'), for the lowest part of the gallbladder to be dissected free from the cystic plate ('liver visible') and for there to be only two structures entering the gallbladder ('2 structures').

REFERENCES:
- [Background] Yamazaki M, Ikeda Y, Ishikawa M, Inagaki C, Tanaka C. [Inhibition of harmaline induced tremor by L-threo-3, 4-dihydroxyphenylserine, an L-norepinephrine precursor]. Nihon Yakurigaku Zasshi. 1976 Apr;72(3):363-9. doi: 10.1254/fpj.72.363. Japanese. PMID 986992
- [Background] Rohner TJ, Hannigan JD, Sanford EJ. Altered in vitro adrenergic responses of dog detrusor msucle after chronic bladder outlet obstruction. Urology. 1978 Apr;11(4):357-61. doi: 10.1016/0090-4295(78)90231-5. PMID 208213
- [Background] Hoffmann MK, Green S, Old LJ, Oettgen HF. Serum containing endotoxin-induced tumour necrosis factor substitutes for helper T cells. Nature. 1976 Sep 30;263(5576):416-7. doi: 10.1038/263416a0. No abstract available. PMID 787802
- [Background] Ditta G, Soderberg K, Scheffler IE. Chinese hamster cell mutant with defective mitochondrial protein synthesis. Nature. 1977 Jul 7;268(5615):64-7. doi: 10.1038/268064a0. No abstract available. PMID 196202
- [Background] Price P. Monitoring response to treatment in the development of anticancer drugs using PET. Nucl Med Biol. 2000 Oct;27(7):691. doi: 10.1016/s0969-8051(00)00140-2. No abstract available. PMID 11091114
- [Background] Price NM. Electron beam therapy. Its effect on eccrine gland function in mycosis fungoides patients. Arch Dermatol. 1979 Sep;115(9):1068-70. doi: 10.1001/archderm.115.9.1068. PMID 114119
- [Background] Carp H, Janoff A. Possible mechanisms of emphysema in smokers. In vitro suppression of serum elastase-inhibitory capacity by fresh cigarette smoke and its prevention by antioxidants. Am Rev Respir Dis. 1978 Sep;118(3):617-21. doi: 10.1164/arrd.1978.118.3.617. PMID 101105